CLINICAL TRIAL: NCT01945502
Title: The Effectiveness of Three Different Nasopharyngeal Packing on the Prevention of Postoperative Nausea- Vomiting and Postoperative Throat Pain in Rhinologic Surgery.
Brief Title: Nasopharyngeal Packing and Rhinologic Surgery.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Basak Ceyda MECO (Other)
Responsible Party: Sponsor-Investigator, Basak Ceyda MECO, MD, DESA, Ankara University
Organization: Ankara University (Other)
Other Study IDs: 11-434-13
Record Dates: First submitted 2013-09-16; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Nasal Surgery; Tampons; PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- nasal packing with dry packs
- nasal packing with wet packs
- nasal packing with Benzidamin-Clorhexsidin damped packs
- no nasal packing

SUMMARY:
The purpose of this study is to assess the efficacy of three different pharyngeal packing during routine rhinologic surgery in the prevention of postoperative nausea and vomiting, and to evaluate the influence of pharyngeal packing on postoperative throat pain.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old adult patient
* nasal and/or paranasal sinus surgeries
* general anesthesia

Exclusion Criteria:

* patients submitted to another intervention at the same time (adenoidectomy, tonsillectomy)
* patients with a serious systemic disease (acquired immunodeficiency syndrome,leukemia, lymphoma, or other neoplasias under chemotherapy treatment)
* patients presenting contraindications for using nonsteroid anti-inflammatory drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients (18-60 years) scheduled for routine nasal and/or paranasal sinus surgeries in Ankara Univerity Faculty of Medicine, ETN operating rooms were recruited into this study.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative nausea vomiting | 3 months
sore throat | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Medicine ENT operating rooms, Ankara, Turkey (Türkiye)